CLINICAL TRIAL: NCT02133950
Title: A Single Centre Randomised Controlled Study Into the Segmentation of Preimplantation Genetic Diagnosis (PGD) Treatment by Comparing Cumulative Pregnancy Rates Following Cryopreservation of All Genetically Transferable Embryos After PGD, Compared to Fresh Embryo Transfer Cumulative With Frozen Embryo Transfer of Genetically Transferable Embryos.
Brief Title: Efficacy Study of Segmentation of PGD Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, VERPOEST WILLEM, professor dr, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.U.N. 143201420647
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Clinical Pregnancy; Live Birth
Keywords: preimplantation genetic diagnosis; cryopreservation; pregnancy
MeSH Terms: interventions — Prostaglandins D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- freeze all embryos following PGD (Experimental): no fresh embryo transfer; elective cryopreservation of all embryos after PGD
  Interventions: Procedure: elective cryopreservation of available embryos after PGD
- elective fresh embryo transfer (Active Comparator)
  Interventions: Procedure: PGD and elective fresh embryo transfer plus cryopreservation of supernumerary available embryos after PGD

INTERVENTIONS:
Procedure: elective cryopreservation of available embryos after PGD — no elective fresh embryo transfer; freeze all
  Other Names: freeze all embryos
  Arms: freeze all embryos following PGD
Procedure: PGD and elective fresh embryo transfer plus cryopreservation of supernumerary available embryos after PGD — PGD and elective fresh embryo transfer plus cryopreservation of supernumerary available embryos after PGD
  Other Names: fresh ET
  Arms: elective fresh embryo transfer

SUMMARY:
A single centre observational study into the segmentation of preimplantation genetic diagnosis (PGD) treatment by comparing cumulative pregnancy rates following cryopreservation of all genetically transferable embryos after PGD, compared to fresh embryo transfer cumulative with frozen embryo transfer of genetically transferable embryos.The primary aim of the study is to assess the feasibility and effectiveness of segmentation in terms of pregnancy rates. The secondary aim is to assess the logistic advantage of segmentation in PGD cycles.

Experimental questions

1. Is the cumulative live birth rate rate of a single PGD treatment when all genetically transferable embryos are cryopreserved by vitrification prior to consecutive in utero transfer in unstimulated cycles, superior to PGD treatment with fresh embryo transfer cumulative with transfer of supernumerary cryopreserved embryos?
2. Does the technique of segmentation allow better planning of DNA amplification and genetic analysis?

Design The proposed design is a pragmatic, prospective randomised controlled trial

ELIGIBILITY:
Inclusion Criteria:

* 1st, 2nd or 3rd cycle of PGD in which embryo transfer was performed
* Indications for PGD: monogenic indications and X-linked disorders with a 25-50% risk of transmission and that are not associated with reduced ovarian response
* Normal ultrasound scan, i.e. presence of both ovaries, without evidence of abnormality within 6 months prior to randomisation.
* Regular menstrual cycles of 21-35 days, presumed to be ovulatory.

Exclusion Criteria:

* POLYCYSTIC OVARIAN SYNDROME (Rotterdam criteria *)

  * At least two of the following three features: (i) Oligo- and/or anovulation (ii) Clinical and/or biochemical signs of hyperandrogenism (iii) Polycystic ovaries and exclusion of other aetiologies (congenital adrenal hyperplasias, androgen-secreting tumours, Cushing's syndrome)
* Poor responders (Bologna criteria **)

  * * At least two of the following three features: (i) Advanced maternal age (≥40 years) or any other risk factor for poor ovarian response (POR); (ii) A previous POR (≤3 oocytes with a conventional stimulation protocol); (iii) An abnormal ovarian reserve test (i.e. antral follicle count (AFC) 5-7 follicles, or anti-Mullerian hormone (AMH) 0.5-1.1 ng/ml).
* Endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney)
* anticipated high response: AMH >5.0 ng/ml or AFC >20
* Endometriosis ≥ grade 3
* Age > 40 years and 364 days

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth rate of a single PGD treatment | 1 year
  cumulative LBR

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Reproductive Medicine UZ Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543